CLINICAL TRIAL: NCT01387984
Title: Association Study of the Plasma Concentration of YKL-40 and Vascular Complications in Patients With Type 2 Diabetes
Brief Title: YKL-40 and Complications in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chih-Hung Lin, MD, National Taiwan University Hospital Yun-Lin Branch
Other Study IDs: 201002053R
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Diabetic complications; YKL-40
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 diabetes mellitus

SUMMARY:
In this study, the investigators plan to establish the relationship between plasma concentration of YKL-40 with various vascular complications in the patients of type 2 diabetes.

DETAILED DESCRIPTION:
It is well recognized now that diabetes mellitus is a systemic vasculopathy and causes various micro- and macrovascular complications. Vascular damage and endothelium dysfunction in diabetes mellitus involve a chronic inflammatory process via a complicated mechanism.

YKL-40 is a 40 kD lectin molecule. It is secreted by various cells, including macrophages, vascular smooth muscle cells and giant cells, and the level of YKL-40 is found elevated in both acute (eg. infection) and chronic (eg. rheumatoid arthritis, systemic lupus erythematosus or cirrhosis of the liver) inflammatory processes. The plasma concentration of YKL-40 is elevated in the patients of type 2 diabetes mellitus compared with non-diabetic controls, and is associated with insulin resistance, fasting plasma glucose and plasma IL-6 concentrations. Furthermore, the concentration of YKL-40 is elevated and is associated with the severity of albuminuria in the patients of type 1 diabetes.

The objective of this study is to establish the relationship between plasma concentration of YKL-40 with various vascular complications in the patients of type 2 diabetes, and to evaluate its potential as a biomarker for the vascular diabetic complications in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Clear consciousness
* type 2 diabetic patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The type 2 diabetic patient who receives follow-up at NTUH diabetics caring network
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2010-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Lin, M.D., Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital Yun-Lin Branch, Douliu City, Yunlin County, Taiwan